CLINICAL TRIAL: NCT04773197
Title: Evaluating a Tailored Cognitive Behavioral Therapy for Adolescent and Young Adult Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2019.159; HUM00165949 (Other: University of Michigan)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Depression, Anxiety; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a three-arm, prospective randomized controlled trial with participants being randomly assigned into one of the three groups: (1) coach-assisted BtB intervention (treatment condition 1), (2) coach-assisted animated EMW (treatment condition 2), and (3) standard BtB (control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coach-assisted C-CBT with BtB (Experimental): Participants will receive coach- assisted Beating the Blues (BtB), a C- CBT program, which contains 8 weekly sessions. A coach will provide between session support throughout the 8 sessions.
  Interventions: Behavioral: Beating the Blues (BtB); Behavioral: Coaching
- Coach-assisted animated C-CBT with EMW (Active Comparator): Participants will receive coach- assisted Entertain Me Well (EMW), an animated C-CBT program, which contains 8 weekly sessions. A coach will provide between session support throughout the 8 sessions.
  Interventions: Behavioral: Entertain Me Well (EMW); Behavioral: Coaching
- Standard stand-alone C-CBT with BtB (Active Comparator): Participants will use the stand-alone BtB for 8 weekly sessions, without coach assistance.
  Interventions: Behavioral: Beating the Blues (BtB)

INTERVENTIONS:
Behavioral: Beating the Blues (BtB) — Beating the Blues (BtB) is a C-CBT intervention with 8 weekly sessions to be completed within 10 weeks.
  Arms: Coach-assisted C-CBT with BtB; Standard stand-alone C-CBT with BtB
Behavioral: Entertain Me Well (EMW) — Entertain Me Well (EMW) is is a C-CBT intervention with 8 weekly sessions to be completed within 10 weeks.
  Arms: Coach-assisted animated C-CBT with EMW
Behavioral: Coaching — A coach will spend approximately 5-10 minutes after each session with the patient to link the C-CBT content with patient's disease specific experiences and to motivate them to continue the program. They will also spend approximately 5 minutes between sessions to motivate a patient to complete assignments and to remind them about starting the next session on time.
  Arms: Coach-assisted C-CBT with BtB; Coach-assisted animated C-CBT with EMW

SUMMARY:
This project's overall goal is to test the feasibility, acceptability and efficacy of two coach-assisted, computer-based, cognitive- behavioral therapy (C-CBT) interventions in treating depression and anxiety in adolescent and young adult cancer survivors. The two coach-assisted interventions will be compared to the standard C-CBT intervention.

DETAILED DESCRIPTION:
This will be a three-arm randomized controlled trial with two treatment arms and one control arm. Participants in the first treatment arm will receive a coach-assisted C-CBT intervention called "Beating the Blues" (BtB). A second treatment arm will receive a coach-assisted, animated C-CBT intervention called "Entertain Me Well" (EMW). Both treatment arms will have 8 weekly sessions that contain core components of CBT. A coach will provide between-session support throughout the 8 sessions. The control arm will use the standard care of BtB without coach assistance.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor, either receiving active treatment or completed cancer treatment
* Experiencing depression and anxiety as measured by PHQ-9 or GAD-7

Exclusion Criteria:

* Severe medical or mental condition (e.g. suicidal ideation)
* Medical condition that prevents patients from operating a computer or tablet
* Receiving end-of-life care

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Rate of C-CBT completion | 10 weeks
  Percentage of participants in each arm who complete at least 6 out of 8 sessions, as measured by online service usage data.
Percentage of participants who confirm acceptability of the intervention during interviews | 10 weeks
  Participants will be interviewed about their perceptions regarding the delivery format, treatment content, and other treatment related factors. Qualitative interviews will be transcribed by research staff and coded using thematic content analysis and axial coding. Qualitative data will be reviewed iteratively until saturation is reached, that is when no new information seems to emerge during coding. Emergence or non-emergence of acceptability theme will be assessed. Findings will be descriptive and will include the percentage of participants who confirm acceptability.

SECONDARY OUTCOMES:
Change in level of depression from baseline to end of intervention | 10 weeks
  The Patient Health Questionnaire, 9 -item (PHQ-9) is a validated brief measure of depression. Participants will answer the questionnaire at their baseline assessment, at the beginning of each session, and at their post-intervention assessment.
Change in level of anxiety from baseline to end of intervention | 10 weeks
  The Generalized Anxiety Disorder, 7-item (GAD-7) is a validated brief measure of anxiety. Participants will answer the questionnaire at their baseline assessment and at their post-intervention assessment.
Change in level of distress from baseline to end of intervention | 10 weeks
  The Brief Symptom Inventory, 18-item (BSI-18) is a validated distress screening tool especially for cancer patients. Participants will answer the questionnaire at their baseline assessment and at their post-intervention assessment.
Change in level of self-efficacy from baseline to end of intervention | 10 weeks
  The PROMIS Self-Efficacy for Managing Chronic Conditions (PROMIS SM Scale) is a 28-item validated tool to assess patients' self-efficacy in managing their chronic condition symptoms.
Change in level of involvement and participation in health care from baseline to end of intervention | 10 weeks
  The Patient Activation Measure (PAM) is a 13-item validated tool to evaluate patients' involvement and participation in their health care. Participants will answer the questionnaire at their baseline assessment and at their post-intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Anao Zhang, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No